CLINICAL TRIAL: NCT02373319
Title: Validity and Effectiveness of a Method for Self-screening of Cardiovascular Risk
Brief Title: Self-screening of Cardiovascular Risk
Acronym: ACRISC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Maria Grau, MD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 5815/I
Record Dates: First submitted 2015-02-20; First posted 2015-02-27 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Risk Factor, Cardiovascular
Keywords: Cardiovascular risk; Cholesterol; Hypertension; Diabetes; Smoking; Preventive Medicine; Epidemiology; Public Health; Diet; Physical Activity
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Smoking; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CV-screening-1 plus personalized (Experimental): Cardiovascular risk screening supervised by health professional - 15 minutes wash-out - Self-screening of cardiovascular risk; Communication of personalized recommendations according to the health exam results for the control of cardiovascular risk factors
  Interventions: Behavioral: CV-screening-1 plus personalized
- CV-screening-2 plus personalized (Experimental): Self-screening of cardiovascular risk - 15 minutes wash-out - Cardiovascular risk screening supervised by health professional; Communication of personalized recommendations according to the health exam results for the control of cardiovascular risk factors
  Interventions: Behavioral: CV-screening-2 plus personalized
- CV-screening-1 plus standard (Active Comparator): Cardiovascular risk screening supervised by health professional - 15 minutes wash-out - Self-screening of cardiovascular risk; Standard communication of the health exam results
  Interventions: Behavioral: CV-screening-1 plus standard
- CV-screening-2 plus standard (Active Comparator): Self-screening of cardiovascular risk - 15 minutes wash-out - Cardiovascular risk screening supervised by health professional; Standard communication of the health exam results
  Interventions: Behavioral: CV-screening-2 plus standard

INTERVENTIONS:
Behavioral: CV-screening-1 plus personalized — Cardiovascular risk screening supervised by health professional - 15 minutes wash-out - Self-screening of cardiovascular risk; Communication of personalized recommendations according to the health exam results for the control of cardiovascular risk factors
  Arms: CV-screening-1 plus personalized
Behavioral: CV-screening-2 plus personalized — Self-screening of cardiovascular risk - 15 minutes wash-out - Cardiovascular risk screening supervised by health professional; Communication of personalized recommendations according to the health exam results for the control of cardiovascular risk factors
  Arms: CV-screening-2 plus personalized
Behavioral: CV-screening-1 plus standard — Cardiovascular risk screening supervised by health professional - 15 minutes wash-out - Self-screening of cardiovascular risk; Standard communication of the health exam results
  Arms: CV-screening-1 plus standard
Behavioral: CV-screening-2 plus standard — Self-screening of cardiovascular risk - 15 minutes wash-out - Cardiovascular risk screening supervised by health professional; Standard communication of the health exam results
  Arms: CV-screening-2 plus standard

SUMMARY:
The aims of this study are (1) to validate a self-screening method for cardiovascular (CV) risk that does not require the supervision of a health professional (including self-measurement of blood pressure, lipid profile evaluated by dry chemistry, and self-administered questionnaires on sex, age, diabetes, and tobacco consumption). (2) From these data, the investigators will generate personalized recommendations based on the best available evidence. The investigators will also analyze whether this innovative approach improves adherence to preventive recommendations for cardiovascular and other chronic diseases.

DETAILED DESCRIPTION:
Primary prevention activities based on some admittedly blunt screening instruments such as cardiovascular (CV) risk functions must be addressed to the whole population, prioritizing certain sectors of the population. However, the main limitation of current risk screening procedures is related to the natural history of cardiovascular disease, whose expression depends on the cumulative exposure to cardiovascular risk factors throughout a person's lifetime. Early prevention of cardiovascular disease is key to reduce this cumulative risk, thereby reducing the incidence of cardiovascular events.

The objectives of this study are (1) to validate a self-screening method for cardiovascular risk that does not require the supervision of a health professional (including self-measurement of blood pressure, lipid profile evaluated by dry chemistry, and self-administered questionnaires on sex, age, diabetes, and tobacco consumption). (2) From these data, the investigators will generate personalized recommendations based on the best available evidence. The investigators will also analyze whether this innovative approach improves adherence to preventive recommendations for cardiovascular and other chronic diseases.

Cardiovascular risk measured with the self-screening method will be compared with the gold standard (cardiovascular risk supervised by health professional). Participants will be randomly assigned to the intervention (communication of cardiovascular risk and recommendation of personalized preventive actions) or control groups (communication of cardiovascular risk). Subjects will be reexamined one year after recruitment for assessing adherence to the preventive recommendations in terms of improvement in the control of cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Understand and accept the study's procedures and sign an informed consent form
* Inhabitants of Girona (Gerona, Spain) and the metropolitan area

Exclusion Criteria:

* History of cardiovascular disease
* Individuals with terminal disease

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 960 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Pre-post changes in blood lipid levels | [Time frame: From baseline to 12 months after the intervention]
  Pre-post changes in mean levels of blood lipid levels (total, HDL and LDL cholesterol). Blood samples will be obtained at baseline and 12 months after the intervention.

SECONDARY OUTCOMES:
Pre-post changes in controlled blood lipid levels | From baseline to 12 months after the intervention
  Pre-post changes in the percentage of individuals with controlled blood lipid levels according to the most updated European Clinical Practice Guidelines (total, HDL and LDL cholesterol). Blood samples will be obtained at baseline and 12 months after the intervention.
Pre-post changes in controlled blood pressure | From baseline to 12 months after the intervention
  Pre-post changes in the percentage of individuals with controlled systolic and diastolic blood pressure levels (140 and 90 mmHg, respectively). Measures will be obtained at baseline and 12 months after the intervention
Pre-post changes in controlled body mass index | From baseline to 12 months after the intervention
  Pre-post changes in the percentage of individuals with body mass index below 25 kg/m2. Measures will be obtained at baseline and 12 months after the intervention.
Pre-post differences in smoking status | From baseline to 12 months after the intervention
  Pre-post changes in the percentage of smokers. Smoking status will be assessed at baseline and 12 months after the intervention
Mean difference between two methods of cardiovascular risk estimation | From baseline to 30 minutes
  Comparison of cardiovascular risk estimates by two methods (Screening of cardiovascular risk supervised by health professional (Gold Standard) - self-screening of cardiovascular risk). Measures with each method will be taken 30 minutes apart after a wash-out period
Pre-post changes in blood pressure | From baseline to 12 months after the intervention
  Pre-post changes in mean levels of systolic and diastolic blood pressure. Measures will be obtained at baseline and 12 months after the intervention.
Pre-post changes in body mass index | From baseline to 12 months after the intervention
  Pre-post changes in mean levels of systolic and diastolic blood pressure. Measures will be obtained at baseline and 12 months after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Grau, MD, PhD, MPH, Principal Investigator — IMIM; Jaume Marrugat, MD, PhD, Study Director — IMIM
Locations (1):
- Unitat de Suport a la Recerca de Girona IDIAP Jordi Gol, Girona, Spain

REFERENCES:
- [Background] Anderson KM, Odell PM, Wilson PW, Kannel WB. Cardiovascular disease risk profiles. Am Heart J. 1991 Jan;121(1 Pt 2):293-8. doi: 10.1016/0002-8703(91)90861-b. PMID 1985385
- [Background] Grau M, Subirana I, Elosua R, Solanas P, Ramos R, Masia R, Cordon F, Sala J, Juvinya D, Cerezo C, Fito M, Vila J, Covas MI, Marrugat J. Trends in cardiovascular risk factor prevalence (1995-2000-2005) in northeastern Spain. Eur J Cardiovasc Prev Rehabil. 2007 Oct;14(5):653-9. doi: 10.1097/HJR.0b013e3281764429. PMID 17925624
- [Background] Kahn R, Robertson RM, Smith R, Eddy D. The impact of prevention on reducing the burden of cardiovascular disease. Circulation. 2008 Jul 29;118(5):576-85. doi: 10.1161/CIRCULATIONAHA.108.190186. Epub 2008 Jul 7. PMID 18606915
- [Background] Kodama S, Saito K, Tanaka S, Maki M, Yachi Y, Asumi M, Sugawara A, Totsuka K, Shimano H, Ohashi Y, Yamada N, Sone H. Cardiorespiratory fitness as a quantitative predictor of all-cause mortality and cardiovascular events in healthy men and women: a meta-analysis. JAMA. 2009 May 20;301(19):2024-35. doi: 10.1001/jama.2009.681. PMID 19454641
- [Background] Marrugat J, Subirana I, Comin E, Cabezas C, Vila J, Elosua R, Nam BH, Ramos R, Sala J, Solanas P, Cordon F, Gene-Badia J, D'Agostino RB; VERIFICA Investigators. Validity of an adaptation of the Framingham cardiovascular risk function: the VERIFICA Study. J Epidemiol Community Health. 2007 Jan;61(1):40-7. doi: 10.1136/jech.2005.038505. PMID 17183014
- [Background] Yusuf S, Hawken S, Ounpuu S, Dans T, Avezum A, Lanas F, McQueen M, Budaj A, Pais P, Varigos J, Lisheng L; INTERHEART Study Investigators. Effect of potentially modifiable risk factors associated with myocardial infarction in 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):937-52. doi: 10.1016/S0140-6736(04)17018-9. PMID 15364185
- [Derived] Barroso M, Zomeno MD, Diaz JL, Perez S, Marti-Lluch R, Cordon F, Ramos R, Cabezas C, Salvador G, Castell C, Schroder H, Grau M. Efficacy of tailored recommendations to promote healthy lifestyles: a post hoc analysis of a randomized controlled trial. Transl Behav Med. 2021 Aug 13;11(8):1548-1557. doi: 10.1093/tbm/ibab035. PMID 33837787
- [Derived] Barroso M, Perez-Fernandez S, Vila MM, Zomeno MD, Marti-Lluch R, Cordon F, Ramos R, Elosua R, Degano IR, Fito M, Cabezas C, Salvador G, Castell C, Grau M. Validity of a method for the self-screening of cardiovascular risk. Clin Epidemiol. 2018 May 10;10:549-560. doi: 10.2147/CLEP.S158358. eCollection 2018. PMID 29785141